CLINICAL TRIAL: NCT05819450
Title: Sonography-Guided Volumetric Rejuvenation on Dorsal Hands: A Split-Hand Randomized Controlled Trial
Brief Title: Sonography-Guided Volumetric Rejuvenation on Dorsal Hands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Teng Hung, Consultant Fellow, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101547B0
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Ultrasound; Injection Site
Keywords: Cosmetic; Volumetric rejuvenation; Filler; Dorsal hand; Ultrasound

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonography-guided hand (Experimental): One hand of the participant will be treated with sonography-guided filler injection in random
  Interventions: Procedure: Volumetric rejuvenation
- Blinded injected hand (No Intervention): One hand of the participant will be treated with filler injection by physician's experience without sonography-guidance in random

INTERVENTIONS:
Procedure: Volumetric rejuvenation — Volumetric Rejuvenation with FDA-approved fillers on the skin of the dorsal hands
  Arms: Sonography-guided hand

SUMMARY:
The goal of this randomized controlled study is to guide volumetric rejuvenation on dorsal hands with the maximal aesthetic appearance. The main questions it aims to answer are:

* Which fatty layer(s) is/are the most suitable for filler injection?
* Is it feasible to make precise filler injections with sonography guidance? Participants will receive sonography-guided injection on the one hand and another with blinded injection.

DETAILED DESCRIPTION:
In our previous study, volumetric fat loss was noted in the 3 fatty laminae of dorsal hands during aging; the dorsal intermediate lamina (DIL) showed the greatest progressive fat loss after the age of 30. Volumetric rejuvenation of the 3 laminae may result in the most aesthetic appearance, especially in women. It is necessary to develop precise rejuvenation therapies according to the aging process of the dorsum of the hands that will yield the most aesthetic appearance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aging changes on the dorsal hands
* Aged ≥18 years

Exclusion Criteria:

* History of severe hand dermatitis
* History of rheumatic arthritis
* History of major hand trauma
* History of limb edema
* History of recent significant weight changes
* History of previous filler injection to the dorsal hands
* History of intravenous catheter insertion and hemodialysis via the forearms or hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Aesthetic improvement | Day 0, 30, 180 follow up
  5-point global aesthetic improvement scales scoring (Min:1; Max:5)

SECONDARY OUTCOMES:
Thickness of the fatty laer | Day 0, 30, 180 follow up
  Thickness of the dorsal superficial lamina (DSL) and dorsal intermediate lamina (DIL)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Teng Hung, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Ocean Clinic Marbella, Marbella, Spain
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No